CLINICAL TRIAL: NCT02461979
Title: The Role of the Vitamin D Receptor Gene Polymorphisms in Hepatocarcinogenesis in Cirrhotic Patients Infected With Chronic Hepatitis C Virus
Brief Title: The Role of the Vitamin D Receptor Gene Polymorphisms in Hepatocarcinogenesis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sherief Abd-Elsalam (Other)
Collaborators: Tanta University (Other)
Responsible Party: Sponsor-Investigator, Sherief Abd-Elsalam, sponsor investigator, Tanta University
Organization: Tanta University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: liver cancer
Record Dates: First submitted 2015-05-31; First posted 2015-06-03 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Hepatocellular carcinoma (HCC) (Other): The VDR genotype in 20 HCV cirrhotic patient with HCC
  Interventions: Other: The VDR genotype
- Liver cirrhosis (Other): The VDR genotype in 20 HCV cirrhotic patient without HCC
  Interventions: Other: The VDR genotype
- Control group (Other): The The VDR genotype in 10 healthy individuals as control
  Interventions: Other: The VDR genotype

INTERVENTIONS:
Other: The VDR genotype — The VDR genotype will determined by polymerase chain reaction (PCR) amplication and restriction length fragment polymorphisms.

SUMMARY:
Previous data have suggested that vitamin D levels may influence cancer development. In particular, several single nucleotide polymorphisms have been described in the Vitamin D receptor( VDR gene), and some polymorphisms are associated with tumor occurrence. For instance, VDR polymorphisms have been related to cancers of the breast, prostate, skin, colon-rectum, bladder and kidney, although with conflicting observations . VDR polymorphisms have also been investigated in the context of some chronic liver diseases, such as chronic hepatitis B, primary biliary cirrhosis and autoimmune hepatitis . In a recent published study, VDR polymorphism may be used as a molecular marker to predict the risk and to evaluate the disease severity of HCC in patients with chronic hepatitis B.

A significant association of VDR (ApaI) polymorphism with the development of HCC in chronic HCV infection may help to identify those who are at high risk of developing HCC.

DETAILED DESCRIPTION:
Hepatitis C virus (HCV) infection is one of the major public health problems worldwide . Chronic HCV infection is characterized by a high rate of progression to fibrosis, chronic hepatitis, leading to cirrhosis and ultimately to hepatocellular carcinoma (HCC). Early detection is critically important because the most effective treatment for HCC is surgical resection or ablation therapy when the tumour is small. On the other hand, genetic factors can also contribute, particularly gene polymorphisms of inflammatory cytokines and growth factor ligands and receptors . Vitamin D is involved in the metabolism of skeleton as a systemic hormone but also has important roles in the regulation of host immune responses, fibrogenesis and development of cancer through vitamin D receptor (VDR). Previous data have suggested that vitamin D levels may influence cancer development. In particular, several single nucleotide polymorphisms have been described in the VDR gene, and some polymorphisms are associated with tumor occurrence. For instance, VDR polymorphisms have been related to cancers of the breast, prostate, skin, colon-rectum, bladder and kidney, although with conflicting observations. VDR polymorphisms have also been investigated in the context of some chronic liver diseases, such as chronic hepatitis B, primary biliary cirrhosis and autoimmune hepatitis . In a recent published study, VDR polymorphism may be used as a molecular marker to predict the risk and to evaluate the disease severity of HCC in patients with chronic hepatitis B.

A significant association of VDR ApaI polymorphism with the development of HCC in chronic HCV infection may help to identify those who are at high risk of developing HCC.

ELIGIBILITY:
Inclusion Criteria:

* Hcv cirrhotic patient with and without Hcc

Exclusion Criteria:

* Malignancy other than HCC
* Co-infection with Hepatitis B virus (HBV) and Human immunodeficiency virus (HIV)
* Cirrhosis is due to causes other than chronic hepatitis C

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-02; Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
number of HCC patients with abnormal (APAL) VDR polymorphism | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Fathia Asal, Prof, Principal Investigator — hepatology dept-Tanta; Amal El Bendary, Professor, Study Director — Clinicalpathology dept-Tanta; WALAA Elkhalawany, lecturer, Study Director — hepatology dept-Tanta; Sherief abd-elsalm, lecturer, Study Chair — hepatology dept-Tanta; Basma Shetaa, physician, Study Chair — Tanta University
Locations (1):
- Tanta university - faculty of medicine, Tanta, Elgharbia, Egypt

IPD SHARING:
Plan to Share IPD: No